CLINICAL TRIAL: NCT02931630
Title: The Effect of Whey Protein and Dietary Fibers on Risk Markers of the Metabolic Syndrome and Bone Health
Acronym: MERITS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other); Rigshospitalet, Denmark (Other); University of California, Davis (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Søren Gregersen, Chief physician, associate professor, ph.d., Aarhus University Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: MERITS
Record Dates: First submitted 2016-08-19; First posted 2016-10-13 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Abdominal Obesity; Metabolic Syndrome; Type 2 Diabetes; Cardiovascular Disease
Keywords: Whey protein; Dietary fibers; Wheat bran; Arabinoxylan; Postprandial lipaemia; Body composition; Blood pressure; Metabolic rate; Insulin sensitivity; Metabolic syndrome
MeSH Terms: conditions — Obesity, Abdominal; Metabolic Syndrome; Diabetes Mellitus, Type 2; Cardiovascular Diseases; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- HP/HF (Experimental): Whey protein powder / High fiber bread
  Interventions: Other: Whey protein powder; Other: High fiber bread
- HP/LF (Experimental): Whey protein powder / Low fiber bread
  Interventions: Other: Maltodextrin powder; Other: Low fiber bread
- LP/HF (Experimental): Maltodextrin powder / High fiber bread
  Interventions: Other: Maltodextrin powder; Other: High fiber bread
- LP/LF (Experimental): Maltodextrin powder / Low fiber bread
  Interventions: Other: Whey protein powder; Other: Low fiber bread

INTERVENTIONS:
Other: Whey protein powder — 60 g of whey protein powder
  Arms: HP/HF; LP/LF
Other: Maltodextrin powder — 60 g of Maltodextrin powder
  Arms: HP/LF; LP/HF
Other: High fiber bread — Wheat bread with high content of dietary fibers (approximately 30 g fibers/day)
  Arms: HP/HF; LP/HF
Other: Low fiber bread — Wheat bread with low content of dietary fibers (approximately 10 g fibers/day)
  Arms: HP/LF; LP/LF

SUMMARY:
The prevalence of overweight and lifestyle related diseases such as cardiovascular disease (CVD) and type 2 diabetes (T2D) is increasing world wide. The metabolic syndrome (MeS) is a condition characterized by abdominal obesity, high blood lipids, high blood pressure and elevated blood sugar. MeS is associated with an increased risk of developing CVD and T2D. Dietary fibers and whey protein have independently shown beneficial effects on several of these risk factors in previous studies. Whey protein is furthermore seen to show positive effects on bone turnover.

The purpose of this trial is to investigate whether an increased intake of dietary fibers and whey protein (separately or combined) over a period of 12 weeks will affect the risk markers of MeS and bone turnover in abdominally obese subjects.

A total of 80 people with abdominal obesity will be included. The design is a randomized, double blinded, controlled dietary intervention trial. Subjects are assigned to one of four experimental groups. Each group are provided with test products containing either high or low whey protein and high or low dietary fibers to replace part of their regular diet. The subjects are instructed in how to incorporate the test products in their habitual diets in order to maintain weight stability.

The primary outcome is postprandial lipaemia (PPL) - an independent risk factor of developing CVD. PPL is estimated by performing a standardized high fat meal test during which postprandial level of triglycerides is measured. The authors hypothesize that a diet of high content of whey protein and high dietary fiber during 12 weeks will induce a reduction in PPL.

DETAILED DESCRIPTION:
Please refer to summary

ELIGIBILITY:
Inclusion Criteria:

* Waist circumference ≥ 80 cm (women)/94 cm (men)
* Age ≥40 years

Exclusion Criteria:

* Significant cardiovascular, renal or endocrine disease
* History of diabetes
* ≥ 3 kg of weight gain or loss within the last 3 months
* Any change in medication within the last month
* Treatment with steroids
* Pregnancy, breastfeeding or planned pregnancy
* Psychiatric history
* Alcohol or drug addiction
* Dietary fiber supplement within the last month

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-06-29 (Actual); Study Completion 2017-06-29 (Actual)

PRIMARY OUTCOMES:
Postprandial triglyceride response | Meal test: -15, 0, 60, 90, 120, 240, 360 min. Performed at baseline and at 12 weeks.
  Postprandial triglyceride response measured as fasting value and incremental Area Under the Curve (iAUC from -15 - 360 min) following a high-fat meal.

SECONDARY OUTCOMES:
24 hours blood pressure (BP) | Performed at baseline and week 12
  Arteriograph 24, TensioMed, Hungary
24 hours augmentation Index (AI) | Performed at baseline and week 12
  Arteriograph 24, TensioMed, Hungary
Respiratory Exchange Ratio | Meal test: -30 and 140 min. Performed at baseline and week 12.
  Measured twice during each meal test by indirect calorimetry (hood)
Body composition | Performed at baseline and week 12
  Dual Energy X-ray Absorptiometry (DEXA) scan: Total body fat percentage, lean mass percentage, gynoid and android fat percentage
Postprandial apolipoprotein B48 response | Meal test: -15, 0, 60, 240, 360 min. Performed at baseline and at 12 weeks.
  Postprandial apolipoprotein response measured as fasting value and incremental Area Under the Curve (iAUC from -15 - 360 min) following a high-fat meal.
Glucose response during high-fat meal test | Meal test: -15, -10, 0, 15, 30, 60, 90, 120, 240, 360 min. Performed at baseline and week 12
  Glucose response measured as fasting value and incremental Area Under the Curve (iAUC from -15 - 360 min) following a high-fat meal.
Insulin response during high-fat meal test | Meal test: -15, -10, 0, 15, 30, 60, 90, 120, 240, 360 min. Performed at baseline and week 12
  Insulin response measured as fasting value and incremental Area Under the Curve (iAUC from -15 - 360 min) following a high-fat meal.
Glucagon response during high-fat meal test | Meal test: -15, -10, 0, 15, 30, 60, 90, 120, 240, 360 min. Performed at baseline and week 12
  Glukagon response measured as fasting value and incremental Area Under the Curve (iAUC from -15 - 360 min) following a high-fat meal.
Glucagon-like peptide 1 (GLP-1) response during high-fat meal test | Meal test: -15, -10, 0, 15, 30, 60, 90, 120, 240, 360 min. Performed at baseline and week 12
  GLP-1 response measured as fasting value and incremental Area Under the Curve (iAUC from -15 - 360
Glucagon-like peptide 2 (GLP-2) response during high-fat meal test | Meal test: -15, -10, 0, 15, 30, 60, 90, 120, 240, 360 min. Performed at baseline and week 12
  GLP-2 response measured as fasting value and incremental Area Under the Curve (iAUC from -15 - 360
Glucose-dependent insulinotropic polypeptide (GIP) response during high-fat meal test | Meal test: -15, -10, 0, 15, 30, 60, 90, 120, 240, 360 min. Performed at baseline and week 12
  GIP response measured as fasting value and incremental Area Under the Curve (iAUC from -15 - 360
Ghrelin response during high-fat meal test | Meal test: -15, -10, 0, 15, 30, 60, 90, 120, 240, 360 min. Performed at baseline and week 12
  Ghrelin response measured as fasting value and incremental Area Under the Curve (iAUC from -15 - 360
Peptide tyrosine tyrosine (PYY) response during high-fat meal test | Meal test: -15, -10, 0, 15, 30, 60, 90, 120, 240, 360 min. Performed at baseline and week 12
  PYY response measured as fasting value and incremental Area Under the Curve (iAUC from -15 - 360
Adiponectin response during high-fat meal test | Meal test: -15, 0, 15, 30, 60, 90, 120, 240, 360 min. Performed at baseline and week 12
  Adiponectin response measured as fasting value and incremental Area Under the Curve (iAUC from -15 - 360)
Non-esterified fatty acids (NEFA) response during high-fat meal test | Meal test: -15, 0, 60, 90, 120, 240, 360 min. Performed at baseline and week 12
  NEFA response measured as fasting value and incremental Area Under the Curve (iAUC from -15 - 360)
Interleukin-6 (IL-6) response during high-fat meal test | Meal test: 0, 15, 30, 60, 90, 120, 240 min. Performed at baseline and week 12
  IL-6 response measured as fasting value and incremental Area Under the Curve (iAUC from 0-240 min)
Monocyte chemoattractant protein 1 (MCP-1) response during high-fat meal test | Meal test: 0, 15, 30, 60, 90, 120, 240 min. Performed at baseline and week 12
  MCP-1 response measured as fasting value and incremental Area Under the Curve (iAUC from 0 - 240 min)
RANTES (CCL5) response during high-fat meal test | Meal test: 0, 15, 30, 60, 90, 120, 240 min. Performed at baseline and week 12
  CCL5 response measured as fasting value and incremental Area Under the Curve (iAUC from 0-240 min)
High-sensitive c-reactive protein (hs-CRP) response during high-fat meal test | Meal test: 0, 15, 30, 60, 90, 120, 240 min. Performed at baseline and week 12
  hs-CRP response measured as fasting value and incremental Area Under the Curve (iAUC from 0-240 min)
Procollagen type 1 N-terminal propeptide (P1NP) response during high-fat meal test | Meal test: 0, 15, 30, 60, 90, 120, 240 min. Performed at baseline and week 12
  P1NP response measured as fasting value and incremental Area Under the Curve (iAUC from 0-240 min)
C-telopeptide (CTX) response during high-fat meal test | Meal test: 0, 15, 30, 60, 90, 120, 240 min. Performed at baseline and week 12
  CTX response measured as fasting value and incremental Area Under the Curve (iAUC from 0-240 min)
Parathyroid hormone (PTH) response during high-fat meal test | Meal test: 0, 15, 30, 90, 240 min. Performed at baseline and week 12
  PTH response measured as fasting value and incremental Area Under the Curve (iAUC from 0-240 min)
Osteoprotegrin response during high-fat meal test | Meal test: 0, 15, 30, 90, 240 min. Performed at baseline and week 12
  Osteoprotegrin response measured as fasting value and incremental Area Under the Curve (iAUC from 0-240 min)
Osteocalcin response during high-fat meal test | Meal test: 0, 15, 30, 90, 240 min. Performed at baseline and week 12
  Osteocalcin response measured as fasting value and incremental Area Under the Curve (iAUC from 0-240 min)
25-dihydroxy vitamin D | Change from week 0 to week 12
  Fasting value measured at baseline and week 12
Phosphate | Change from week 0 to week 12
  Fasting value measured at baseline and week 12
Magnesium | Change from week 0 to week 12
  Fasting value measured at baseline and week 12
Total cholesterol | Change from week 0 to week 12
  Fasting value measured at baseline and week 12
Low density lipoprotein (LDL) | Change from week 0 to week 12
  Fasting value measured at baseline and week 12
High density lipoprotein (HDL) | Change from week 0 to week 12
  Fasting value measured at baseline and week 12
Glucose response during oral glucose tolerance test (OGTT) | OGTT: -15, -10, 0, 30, 60, 90, 120 min. Performed at baseline and week 12
  Glucose measured as incremental Area Under the Curve (iAUC from -15 - 120 min)
Insulin response during oral glucose tolerance test (OGTT) | OGTT: -15, -10, 0, 30, 60, 90, 120 min. Performed at baseline and week 12
  Insulin measured as incremental Area Under the Curve (iAUC from -15 - 120 min)
Glucagon response during oral glucose tolerance test (OGTT) | OGTT: -15, -10, 0, 30, 60, 90, 120 min. Performed at baseline and week 12
  Glucagon measured as incremental Area Under the Curve (iAUC from -15 - 120 min)
Glucagon-like peptide 1 (GLP-1) response during oral glucose tolerance test (OGTT) | OGTT: -15, -10, 0, 30, 60, 90, 120 min. Performed at baseline and week 12
  GLP-1 measured as incremental Area Under the Curve (iAUC from -15 - 120 min)
Glucagon-like peptide 2 (GLP-2) response during oral glucose tolerance test (OGTT) | OGTT: -15, -10, 0, 30, 60, 90, 120 min. Performed at baseline and week 12
  GLP-2 measured as incremental Area Under the Curve (iAUC from -15 - 120 min)
Glucose-dependent insulinotropic polypeptide (GIP) response during oral glucose tolerance test (OGTT) | OGTT: -15, -10, 0, 30, 60, 90, 120 min. Performed at baseline and week 12
  GIP measured as incremental Area Under the Curve (iAUC from -15 - 120 min)
Parathyroid hormone (PTH) response during oral glucose tolerance test (OGTT) | OGTT: 0, 30, 90 min. Performed at baseline and week 12
  PTH measured as incremental Area Under the Curve (iAUC from 0-90 min)
C-telopeptide (CTX) response during oral glucose tolerance test (OGTT) | OGTT: 0, 30, 90 min. Performed at baseline and week 12
  CTX measured as incremental Area Under the Curve (iAUC from 0-90 min)
Procollagen type 1 N-terminal propeptide (P1NP) response during oral glucose tolerance test (OGTT) | OGTT: 0, 30, 90 min. Performed at baseline and week 12
  P1NP measured as incremental Area Under the Curve (iAUC from 0-90 min)
Osteoprotegrin response during oral glucose tolerance test (OGTT) | OGTT: 0, 30, 90 min. Performed at baseline and week 12
  Osteoprotegrin measured as incremental Area Under the Curve (iAUC from 0-90 min)
Osteocalcin response during oral glucose tolerance test (OGTT) | OGTT: 0, 30, 90 min. Performed at baseline and week 12
  Osteocalcin measured as incremental Area Under the Curve (iAUC from 0-90 min)
Waist and hip circumference. | Change from week 0 to week 12
  Waist and hip circumference in cm
Body weight | Change from week 0 to week 12
  Body weight in kg
Body Mass Index | Change from week 0 to week 12
  kg/m2
Adipose tissue gene expression | Change from week 0 to week 12
  Subcutaneous fat tissue biopsy performed at baseline and week 12 for the measurement of changes in genes related to lipid and glucose metabolism and insulin signalling.
Adipose tissue proliferation and differentiation | Change from week 0 to week 12
  Subcutaneous fat tissue biopsy performed at baseline and week 12 for measuring proliferation and differentiation processes of preadipocyte stem cells into mature adipocytes, and to test the effect of diets on expanding the capacity of the subcutaneous adipose tissue to store fat.
Urinary calcium | Change from week 0 to week 12
  Urinary calcium excretion measured in 24-hour urine samples collected at baseline and week 12
Urinary nitrogen | Change from week 0 to week 12
  Urinary nitrogen excretion measured in 24-hour urine samples collected at baseline and week 12
Metabolomics, plasma | OGTT: -15, 30, 60, 90, 120 min. Performed at baseline and week 12.
  Non-targeted metabolomics analysis using Liquid Chromatography - Mass Spectrometry
Metabolomics, urine | 24-hour urine collection performed at baseline and week 12.
  Non-targeted metabolomics analysis using Liquid Chromatography - Mass Spectrometry
Metabolomics, faeces | Collected at baseline and week 12.
  Non-targeted metabolomics analysis using Liquid Chromatography - Mass Spectrometry
Insulin sensitivity during oral glucose tolerance test (OGTT) | OGTT performed at baseline and week 12 (blood sampling at -15, -10, 0, 30, 60, 90, 120 min)
  Homeostasis model assessment - insulin resistance (HOMA-IR) and Matsuda Index calculated based on blood glucose and insulin measurements during OGTT
Appetite assessment during high-fat meal test | Meal test: Questionnaire at -10, 0, 30, 60, 90, 120, 180, 240, 300, 360 min. Performed at baseline and week 12.
  Visual Analog Scale (VAS) electronic questionnaire
Microbiota | Faecal samples collected at baseline and week 12.
  Non-targeted microbiome and metabolome analyses using high-throughput DNA sequencing on Illumina Miseq and Liquid Chromatography - Mass Spectrometry (LC-MS) metabolomics,

CONTACTS AND LOCATIONS:
Overall Officials: Søren Gregersen, MD, ph.d., Principal Investigator — Aarhus University Hospital; Knud Erik B. Knudsen, Professor, Study Chair — Department of Animal Science, University of Aarhus
Locations (1):
- Aarhus University Hospital, Dep. of clinical nutrition research, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fuglsang-Nielsen R, Rakvaag E, Vestergaard P, Hermansen K, Gregersen S, Starup-Linde J. The Effects of 12-Weeks Whey Protein Supplements on Markers of Bone Turnover in Adults With Abdominal Obesity - A Post Hoc Analysis. Front Endocrinol (Lausanne). 2022 Mar 29;13:832897. doi: 10.3389/fendo.2022.832897. eCollection 2022. PMID 35422766